CLINICAL TRIAL: NCT04836520
Title: Single-arm, Single-center, PhaseⅡ Clinical Study of SHR6390 Combined With Anastrozole for Preoperative Treatment of Hormone Receptor Positive and HER2 Negative Early or Locally Advanced Breast Cancer.
Brief Title: SHR6390 Combined With Anastrozole for Preoperative Treatment of Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-NEO-IIT-SHR6390
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR6390+anatrozole (Experimental): Hormone receptor positive, HER2 negative participants will receive SHR6390 in combination with anatrozole before surgery.
  Interventions: Drug: SHR6390+anatrozole

INTERVENTIONS:
Drug: SHR6390+anatrozole — SHR6390 is a novel small molecule inhibitor specifically targeting the CDK4/6 pathway.

SUMMARY:
The study is being conducted to assess effect of SHR6390 combined with anastrozole on proliferation of HR-positive HER2-negative breast cancer tumor cells before surgery.

DETAILED DESCRIPTION:
This is a single-arm, single-center, open-label Phase II clinical study. The purpose of this study was to evaluate the effect of SHR6390 combined with anastrozole on the proliferative activity of HR-positive HER2-negative breast cancer tumor cells before surgery.

ELIGIBILITY:
Inclusion Criteria:

1.Female subjects aged 18 to 75 years old, meet any of the following:

1. Both ovaries have been removed, or the age is ≥60 years old;
2. Age <60 years, natural post-menopausal state (defined as spontaneous menstrual cessation for at least 12 consecutive months without other pathological or physiological reasons), E2 and FSH are at postmenopausal levels;
3. Premenopausal or perimenopausal female subjects must be willing to receive LHRH agonist treatment during the study; 2.T2-T4cN0M0 invasive breast cancer (according to the AJCC 8th edition breast cancer clinical staging guidelines), the tumor must be surgically resectable, the measurable lesion conforms to the RECIST 1.1 standard, and the maximum diameter of the primary tumor has been evaluated by clinical or imaging evaluation ≥ 2cm; 3.Willing to accept biopsy; 4.Luminal A confirmed by immunohistochemistry, ER≥50% and PR≥50%; 5.HER2 negative, defined as immunohistochemical test 0/1+; or FISH test HER2/CEP17 ratio is less than 2.0 or HER2 gene copy number is less than 4; 6.Patients are suitable for neoadjuvant therapy and willing to accept (judged by the investigator); 7.ECOG performance status score 0 or 1; 8.The expected survival period is not less than 12 weeks; 9.Adequate function of major organs； 10.Voluntary participation in the study, signed informed consent, good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Metastases confirmed by imaging or pathology, not including lymph node metastases in the ipsilateral and/or contralateral thoracic region or mediastinum;
2. Inflammatory breast cancer, bilateral breast cancer or DCIS, invasive breast cancer with multiple focal lesions;
3. Previous pathological diagnosis of HER2-positive breast cancer;
4. Suffering from gastrointestinal diseases such as intestinal obstruction, peptic ulcer or active bleeding, which affects the taking and absorption of drugs;
5. Previously treated with radiotherapy, chemotherapy, surgery (not including percutaneous puncture) or molecular targeted treatment;
6. Previously received any CDK4/6 inhibitor drug treatment;
7. Participation in any other clinical trials within 4 weeks of enrollment；
8. Concurrent use of any other Anti-cancer drugs；
9. Other malignancies within 5 years, except cured in-situ of uterine cervix carcinoma , skin basal cell carcinoma and squamous-cell carcinoma;
10. History of heart disease: (1) Arrhythmias requiring medical treatment or clinical significance, (2) Myocardial infarction, (3) Heart failure, (4)Any heart diseases that investigator believes not suitable for this study;
11. History of allergy or hypersensitivity to any of the study drugs or study drug components; history of immunodeficiency including HIV-positive, active hepatitis B/C, other acquired, congenital immunodeficiency disease or history of organ transplantation；
12. A clear history of neurological or mental disorders, including epilepsy or dementia；
13. Pregnant or breastfeeding women. Women of childbearing potential who have a positive pregnancy test or unwilling to use adequate contraception prior to enrollment and for the duration of study participation；
14. According to the investigator's judgment, there is a concomitant disease that seriously endangers the safety of subjects or affects the completion of the study (including but not limited to severe hypertension, severe diabetes, active infection, thyroid disease that cannot be controlled by drugs)；
15. Any condition which in the investigator's opinion makes the subjects unsuitable for the study participation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in Ki67 scores | up to 5 months
  Serial measures of Ki67 (%)
RCB (0-1) after surgery | 5 months
  Rate of Residual Cancer Burden 0-1

SECONDARY OUTCOMES:
Objective response rate (ORR) evaluated by the investigator | 16 weeks
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) according to RECIST 1.1.
tpCR | 5 months
  pCR is defined as the absence of noninvasive tumor residuals in breast and axillary lymph nodes (ypT0/is ypN0) after neoadjuvant therapy.
Safety will be assessed using NCI Common Terminology Criteria for Adverse Events v5.0 (CTCAE) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- TianJin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No